CLINICAL TRIAL: NCT06978023
Title: Clinical Safety, Efficacy and Multiomic Evaluation of a Novel Chinese Medicine Formula in Type 2 Diabetes: Effects on Beta-cell Function and Insulin Resistance
Brief Title: Novel Chinese Medicine Formula for Diabetes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JM_RCT_2024
Record Dates: First submitted 2025-05-01; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; Chinese medicine; insulin; multiomic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JM-LD group (Experimental): Name: JM-LD packed in illumina foil Form: powder dissolved in 250 ml hot water Dosage 13.5 g per packet Frequency: twice daily Duration: 24 weeks
  Interventions: Combination Product: JM-LD
- JM-HD group (Experimental): Name: JM-HD packed in illumina foil Form: powder dissolved in 250 ml hot water Dosage 13.5 g per packet Frequency: twice daily Duration: 24 weeks
  Interventions: Combination Product: JM-HD
- Placebo group (Placebo Comparator): Name: Placebo in illumina foil Form: powder dissolved in 250 ml hot water Dosage 13.5 g per packet Frequency: twice daily Duration: 24 weeks
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: JM-LD — Proprietary formula of extracts of Coptidis Rhizoma, Astragali Radix Lonicerae Japonicae Flos (CAL) plus low dose extract of Ophiopogonis Radix
  Other Names: Jinmai (CAL+ low dose Ophiopogonis Radix)
  Arms: JM-LD group
Combination Product: JM-HD — Proprietary formula of extracts of Coptidis Rhizoma, Astragali Radix, Lonicerae Japonicae Flos (CAL) plus high dose extract of Ophiopogonis Radix
  Other Names: Jinmai (CAL+ high dose Ophiopogonis Radix)
  Arms: JM-HD group
Combination Product: Placebo — Placebo consisting of excipients, coloring and food ingredients to provide a powder mixture of same weight with similar color, texture and odour
  Arms: Placebo group

SUMMARY:
Diabetes is a leading cause of heart disease, stroke, kidney failure, cancer and premature death. One in 10 adults are affected by diabetes. Early control of high blood gluocse prevents progressive deterioration and treatment escalation. People with diabetes have impaired insulin secretion, the only hormone that can lower blood glucose, or resistance to insulin action. There are trillions of microrganisms (tiny living things including bacteria) in the gut that can interact with foods and medicine to alter bodily functions including insulin secretion and its actions. Studies in animals and human suggested that a Traditional Chinese Medicine (TCM) containing a combination of four herbs (Jinmai, abbreviated as JM) reduced blood glucose by increasing insulin secretion accompanied by favorable changes in gut bacteria and expression of genetic information that regulate bodily functions.

In this study, people with type 2 diabetes diagnosed for less than 6 years and not treated with any glucose lowering drugs are assigned randomly to recieve 1) high dose JM (JM-HD) or 2) low dose JM (JM-LD) or 3) look-alike dummy (placebo) given in powder form to be dissolved in water taken twice daily for 24 weeks. We shall compare the abilities of these 3 combination products to lower blood glucose over a 2-hour period after taking a nutritional drink at 0, 12 and 24 weeks. The assigned treatment will then be discontinued for 12 weeks and the test will be repeated to see if improvement is sustained. Samples will be collected at week 0 and 24 (on-treatment) and week 36 (12 weeks off-treament) to compare changes in gut bacteria in faeces and expression of genetic information that make proteins which regulate blood glucose amongst these 3 groups.

DETAILED DESCRIPTION:
People with impaired insulin secretion from the pancreatic beta-cells is the main cause of type 2 diabetes (T2D). This can be demonstrated by measuring insulin secretion following an 75 gram oral glucose tolerance test (OGTT) or a mixed meal tolerance test (MMTT). Other pathophysiological processes underlying diabetes include non-suppression of glucagon from pancreatic alpha-cells with increased fasting blood glucose, abnormal incretin (e.g. glucagon like peptide GLP1) secretion from gut which augment insulin secretion during food intake as well as changes in gut microbiota which can interact with foods and medicine to alter hormonal secretion and metabolic milieu. Obesity, hyperglycaemia and dyslipidemia can alter inflammatory pathways, transcription factors and oxidative stress resulting in further impairment of insulin secretion and its actions. Early attainment of glycemic control can break these vicious cycles, improve glycemic durability and reduce progressive treatment escalation.

Several randomized controlled trials (RCTs) and meta-analyses indicate that TCM containing multiple active components may prevent and control diabetes in human. In animal studies, our group first reported that a combination of extracts from 3 herbs (Coptidis Rhizoma; Astragali Radix; Lonicerae Japonicae Flos, abbreviated as CAL) lowered blood glucose in diabetic rats with sustained improvement in insulin resistance and beta-cell function accompanied by resolution of fatty liver. These effects persisted for weeks or months after treatment discontinuation depending on treatment duration. These improvements were accompanied by changes in gene expression (RNA and microRNA) implicated in energy metabolism. In another animal study, we first reported that extracts from Ophiopogonis (Oph) increased insulin secretion, reduced inflammation and expanded islet mass with lowering of blood glucose.

Based on these mechanistic studies, we designed a proprietary formula consisting of CAL plus Oph (referred as Jinmai, JM). We randomized people with prediabetes to recieve 12-week treatment with 1) CAL only, 2) CAL+Oph low dose (JM-LD), 3) CAL+Oph very low dose (JM-VLD) and 4) consultation with CM practitioners (control), followed by treatment discontinuation for 12 weeks. Amongst these 4 groups, participants treated with JM-LD had signficant reduction in blood glucose and increased insulin secretion during 75 gram OGTT. This effect was sustained after discontinuation of JM-LD for 3 months. Microbiota and RNA analysis indicated that JM-LD caused favorable changes in microbiota and gene expression which correlated with these metabolic changes.

Based on these consistent evidence, we produced a proprietary JM formula consisting of a fixed combination of extracts of CAL with low dose (JM-LD) or high dose extracts of Oph (JM-HD) under good manufacturing practice. The study was approved by the Hong Kong Department of Health for investigational use aimed at registering JM as a novel CM for prevention and treatment of T2D.

Hypothesis:

A 24-week treatment with JM in people with T2D reduce glucose excursion and improve beta-cell function through changes in gut microbiota and gene expression

Study design:

A double-blind, placebo-controlled RCT to assess the efficacy, safety and multiomic effects of JM and its optimal dose in people with early T2D (within 6 years) not treated with glucose lowering drugs.

Intervention:

Randomized in a 1:1:1 ratio to receive 24-week treatment with

1. JM-LD in powder form (13.5 g twice daily) to be dissolved in 250 ml of hot water
2. JM-HD in powder form (13.5 g twice daily) to be dissolved in 250 ml of hot water or
3. matching placebo in powder form (13.5 g twice daily) to be dissolved in 250 ml of hot water followed by treatment discontinuation for 3 months

Primary objective:

To compare changes in glucose excursion during MMTT after 24 week treatment with JM-LD or JM-HD compared to placebo

Secondary objectives:

1. To evaluate the sustained effect of JM on glucose exursion during MMTT 12 weeks after JM discontinuation compared to placebo
2. To compare changes in cardiometabolic risk factors including blood pressure, lipids and body weight and HbA1c as well as insulin secretion and resistance during MMTT after 24 weeks of JM treatment compared to placebo
3. To compare changes in biomarkers and multiomics and their correlations with metabolic changes after 24 weeks of JM treatment compared to placebo

Primary outcome measure:

Between-group difference in area-under-the-curve of plasma glucose (AUC-PG) during MMTT in the JM group versus changes in the placebo group (difference-difference) from week 0 to 24 (on treatment)

Sample size:

In the aforementioned 12-week study of JM versus placebo in people with prediabetes, the mean (SD) of AUC-PG during OGTT in placebo group was 18.9 (1.8) mmol/L/min. The AUC-PG was 1.89 mmol/L/min, i.e. 10% lower in the JM-LD group than the placebo group. Based on a conservative estimation of a superiority margin of 0.945 (5% of mean difference) in favor of JM-HD versus placebo, 45 participants in each arm are needed to achieve an 80% power at one-sided significance level of 5%. Allowing a 20% drop out rate, we shall assign 54 participants to each of 3 groups with a total of 162 participants.

Study site:

The study will be conducted at Ward 3M, Diabetes and Endocrine Research Centre, Prince of Wales Hospital in accordance with Declaration of Helsinki, and Good Clinical Practice (GCP) and Standard Operation Procedures (SOP) stipulated by the CUHK-NTEC Clinical Research Management Office

Significance of the study:

This double-blind placebo-controlled RCT will provide data in support of the beneficial effects of a novel proprietary CM formula (JM) on glycemic excursion in people with early T2D as a therapeutic option. The effects of JM on beta-cell function, insulin resistance, biomarkers, multiomics and gut microbiota will explain the mechanisms underlying the benefits of JM. These data will provide the basis for conduct of large-scale study to examine the effects of JM in the prevention of T2D and its progression to non-communicable diseases.

ELIGIBILITY:
Inclusion criteria:

* Diabetes based on 1) HbA1c≥6.5% OR 2) 75-gram OGTT (fasting PG ≥7 mmol/L or 2-h PG≥11.1 mmol/L) with 2 abnormal values in individuals without symptoms or 1 abnormal value in individuals with symptoms
* HbA1c≤8%
* Age ≥18 years - 70 years (inclusive)
* Body mass index (BMI) ≥18 kg/m2
* Chinese ethnicity
* Duration of T2D (no history of ketosis or continuous requirement of insulin within 12 months of diagnosis) ≤ 6 years
* Not on any glucose lowering drugs for the last 3 months

Exclusion criteria:

* Not willing to participate in the study or adhere to study procedures
* Significant medical history including but not limited to history of cardiovascular disease (stroke, ischaemic heart disease, peripheral vascular disease) within the last 6 months, estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2 and/or liver dysfunction (AST and/or ALT≥1.5 times upper limit of normal)
* History of drug abuse or excessive alcohol intake based on investigator judgment
* Dehydration, diarrhea or vomiting at the time of recruitment
* Individuals with severe infection, in perioperative period or with serious injury at the time of recruitment
* Individuals with blood haemoglobin outside the normal range (male: 13.5-17.5 g/dl and female: 12.0-15.5 g/dl)
* Use of dietary supplements or health products which might affect glucose metabolism or body weight within 1 month before first dose, as judged by the investigator
* Breast feeding, pregnant women or women with plans for pregnancy
* Individuals using warfarin or other medications which may cause herb-drug interactions as judged by the investigator
* Individuals with known G6PD deficiency or known history of herb-drug interactions
* HbA1c >8.0% at screening, treated or untreated
* Use of weight loss drugs currently or within 1 month before first dose
* Use of any glucose lowering drugs
* Previous metabolic surgery
* Known history of thyroid disorders
* History of clinically significant drug hypersensitivity reactions
* Use of any investigational drug within 3 months prior to screening
* Use of any sensitive substrates or organic anion transporter (OAT) 1 or 2, or inhibitors of OAT1 or OAT2 from randomization to the study close out visit (Examples of OAT1 substrates include adefovir, ciprofloxacin, furosemide, tenofovir. Examples of OAT2 substrate include metformin. Examples of OAT1 inhibitors include probenecid. Examples of OAT2 inhibitors include cimetidine, dolutegravir, isavuconazole, ranolazine).
* Use of any OATP1B1 transporter substrates from randomization to the study close out visit (Examples include atorvastatin, lovastatin, pitavastatin, pravastatin, glyburide, paclitaxel, exofenadine, elagolix, docetaxel, bosentan).
* Use of any P-gp substrates or P-gp inhibitors from randomization to the study close out visit (Examples of P-gp substates include digoxin, fexofenadine, dabigatran etexilate, edoxaban. Examples of P-gp inhibitors include amiodarone, clarithromycin, erythromycin, itraconazole, ketoconazole, cobicistat, cyclosporine, dronedarone, lapatinib, lopinavir and ritonavir)
* BP ≥140 mmHg (systolic) or 90 mmHg (diastolic) treated or untreated.
* Any conditions considered unsuitable by the investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Difference-difference in glycemic excursion during MMTT after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in area under the curve of plasma glucose (AUC-PG) during 2-hour MMTT in JM group versus changes in the placebo group

SECONDARY OUTCOMES:
Difference-difference in glycemic excursion during MMTT 12 weeks off JM treatment | From Week-24 to Week-36 (off treatment)
  Between-group difference in AUC-PG during 2-hour MMTT in JM group versus changes in placebo group
Difference-difference in insulin resistance after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in HOMA-IR in the JM group versus changes in placebo group
Difference-difference in beta cell function after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in HOMA-beta in the JM group versus changes in placebo group
Difference-difference in insulin secretion after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in insulinogenic index derived from PG and insulin measured during MMTT in the JM group versus changes in placebo group
Difference-difference in insulin sensitivity after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in quantitative insulin sensitivity check index (QUICKI) derived from PG and insulin measured during MMTT in the JM group versus changes in placebo group
Difference-difference in body mass index (BMI) after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in BMI in JM group versus changes in placebo group
Difference-difference in blood pressure after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in blood pressure in JM group versus changes in placebo group
Difference-difference in non-HDL cholesterol after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in non-HDL cholesteroal in JM group versus changes in placebo group
Difference-difference in HbA1c after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in HbA1c in JM group versus changes in placebo group
Difference-difference in waist circumference after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in waist circumference in JM group versus changes in placebo group
Difference-difference in blood haemoglobin after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in blood haemoglobin in the JM group versus changes in placebo group
Difference-difference in estimated glomerular filtration rate (eGFR) after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in ichanges in eGFR in the JM group versus changes in placebo group
Difference-difference in serum alanine transferase after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in serum alanine transferase in the JM group versus changes in placebo group
Difference-difference in serum alkaline phosphatase after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in ichanges in serum alkaline phosphatase in the JM group versus changes in placebo group
Difference-difference in serum bilirubin after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in serum bilirubin in the JM group versus changes in placebo group
Difference-difference in EQ5D index after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in EQ5D as index of quality of life in the JM group versus changes in the placebo group

OTHER OUTCOMES:
Difference-difference in glucagon like peptide (GLP-1) after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in GLP-1 in the JM group versus changes in the placebo group
Difference-difference in gut microbiome after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in microbiome in the JM group versus changes in the placebo group
Difference-difference in blood RNA expression after 24 weeks of JM treatment | From Week-0 to Week-24
  Between-group difference in changes in RNA expression in the JM group versus changes in the placebo group
Relationships between metabolic and multiomic changes | From Week-0 to Week-24
  Correlations between changes in outcome measures and changes in microbiome and RNA

CONTACTS AND LOCATIONS:
Overall Officials: Juliana CN CHAN, MD, Principal Investigator — CUHK
Locations (1):
- Department of Medicine and Therapeutics, The Chinese University of Hong Kong (CUHK), Ward 3M, Diabetes and Endocrine Research Centre, 3/F Day Treatment Block and Children Wards (Old Block), Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao HL, Sui Y, Qiao CF, Yip KY, Leung RK, Tsui SK, Lee HM, Wong HK, Zhu X, Siu JJ, He L, Guan J, Liu LZ, Xu HX, Tong PC, Chan JC. Sustained antidiabetic effects of a berberine-containing Chinese herbal medicine through regulation of hepatic gene expression. Diabetes. 2012 Apr;61(4):933-43. doi: 10.2337/db11-1164. Epub 2012 Mar 6. PMID 22396199
- [Background] Mao D, Tian XY, Mao D, Hung SW, Wang CC, Lau CBS, Lee HM, Wong CK, Chow E, Ming X, Cao H, Ma RC, Chan PKS, Kong APS, Li JJX, Rutter GA, Tam WH, Chan JCN. A polysaccharide extract from the medicinal plant Maidong inhibits the IKK-NF-kappaB pathway and IL-1beta-induced islet inflammation and increases insulin secretion. J Biol Chem. 2020 Sep 4;295(36):12573-12587. doi: 10.1074/jbc.RA120.014357. Epub 2020 Jun 30. PMID 32605924